CLINICAL TRIAL: NCT06398184
Title: Motor Imagery and Action Observation in Patients With Knee Osteoarthritis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cardenal Herrera University (Other)
Responsible Party: Principal Investigator, Luis Suso, PhD, Cardenal Herrera University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MI1
Record Dates: First submitted 2024-04-23; First posted 2024-05-03 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-04

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise + motor imagery and action observation (Experimental)
  Interventions: Other: Exercise + motor imagery and action observation
- Exercise (Active Comparator)
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise + motor imagery and action observation — A total of 8 sessions of 4 sets of knee extension exercises will be performed. During the breaks between each series, participants will perform a progressive protocol of action observation and motor imagery.
  Arms: Exercise + motor imagery and action observation
Other: Exercise — A total of 8 sessions of 4 sets of knee extension exercises will be performed.
  Arms: Exercise

SUMMARY:
The main objective of this study is to evaluate the effects of an exercise programme combined with motor imagery and action observation, both in the short and long term.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with severe knee OA (according to the clinical and radiographic criteria of the American College of Rheumatology Guidelines)

Exclusion Criteria:

* pain in the contralateral (non-studied) limb (maximum ≥80 of 100 mm on a visual analog scale (VAS) during daily activities),
* undergone another hip or knee joint replacement in the previous year
* any medical condition in which exercise was contraindicated or if they had participated in exercise programs or motor imagery/action observation intervention

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-05-15 (Estimated); Primary Completion 2024-10-15 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Pain intensity (Visual analogue scale) | through study completion, 1 month
  Pain intensity will be measured using a visual analogue scale.
Disability (WOMAC scale) | through study completion, 1 month
  Disability will be measured using WOMAC scale.
Algometry | through study completion, 1 month
  Pressure pain thresholds will be measured by algometry on the affected knee, contralateral knee and epicondyle.